CLINICAL TRIAL: NCT00963053
Title: A Randomised, Double Blind, Placebo Controlled, Multicentre, Cross Over Proof of Concept Study to Investigate the Efficacy and Safety of Pre Emptive Administration of Repeated, Oral Doses of VA111913 TS for the Alleviation of Dysmenorrhoea
Brief Title: VA111913 Dysmenorrhoea Efficacy and Safety Proof of Concept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 913-002
Record Dates: First submitted 2009-08-17; First posted 2009-08-21 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Primary Dysmenorrhea
Keywords: dysmenorrhoea; dysmenorrhea; pain; pre-emptive
MeSH Terms: conditions — Dysmenorrhea; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VA111913 100mg twice daily (Experimental)
  Interventions: Drug: VA111913 TS and placebo
- Starch pill (Placebo Comparator)
  Interventions: Drug: VA111913 TS and placebo

INTERVENTIONS:
Drug: VA111913 TS and placebo — VA111913 TS twice daily for a maximum of 6 days during one menstrual cycle followed by placebo twice daily for up to a maximum of 6 days during a second menstrual cycle in a cross over design

SUMMARY:
The purpose of the study is to investigate how effective VA111913 is at preventing menstrual pain in women with primary dysmenorrhoea.

DETAILED DESCRIPTION:
Dysmenorrhoea is suffered by between 50% and 90% of women of child bearing age. Up to 30% of these women are non-responsive to the currently prescribed therapies. As such it represents an area of unmet medical need. VA111913 inhibits vasopressin-induced contractions of human myometrial strips and human myometrial blood vessels in vitro. By this mechanism, it is anticipated that the pain of dysmenorrhoea, a condition in which myometrial tone and contractions are increased and blood flow to the uterus is decreased compared to normal, may be reduced.

Subjects will be dosed with VA111913 TS and placebo in a cross over design during two consecutive menstrual cycles. They will be dosed for up to a maximum of 6 days, beginning 2 days before the onset of menstruation. Subjects will then assess the menstrual pain, bleeding and amount of analgesia required to treat symptoms during each cycle

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 35 years old
* Not pregnant
* History of primary dysmenorrhoea
* Regular menstrual cycles
* Signed informed consent

Exclusion Criteria:

* Known secondary dysmenorrhoea
* Concomitant use of regular prescription or non prescription medications or herbal remedies
* Any clinically significant medical history or active disease
* Participation in another clinical study in the last 3 months
* Contraindication to chosen rescue medications or allergy to their constituents
* Other protocol defined eligibility criteria may apply

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pain assessed using standard scoring system | 3 months

SECONDARY OUTCOMES:
Safety assessed by laboratory findings, vital signs, ECGs and AEs | 3 months
Assessment of treatment effectiveness | 3 months
Requirement for rescue medication | 3 months
Assessment of menstrual bleeding | 3 months
PK assessments | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David Bell, Principal Investigator — Bio-Kinetic Europe Limited; Stephen E Daniels, Principal Investigator — Premier Research; Vernon Yamashiro, Principal Investigator — Jean Brown Research; Louise Taber, Principal Investigator — Pivotal Research Centers
Locations (4):
- United States (3):
  - Pivotal Research Centers, Peoria, Arizona
  - Premier Research Group, Austin, Texas
  - Jean Brown Research, Salt Lake City, Utah
- Bio-Kinetic Europe Limited, Belfast, United Kingdom